CLINICAL TRIAL: NCT06717685
Title: Comparison of Verapamil With Adenosine After Vagal Maneuvers in Patients Presenting With Paroxysmal Supraventricular Tachycardia (pSVT), in a Tertiary Care Hospital of Lahore, Pakistan
Brief Title: Efficacy of Adenosine as Compared to Verapamil in Paroxysmal Supraventricular Tachycardia (pSVT) Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Rashid Latif Medical College (Other)
Collaborators: Punjab Institute of Cardology (Other); Himmel Pharmaceutical private limited, Pakistan (Unknown)
Responsible Party: Principal Investigator, Arslan Saleem, Biostatistician, Rashid Latif Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PIC001/2024
Record Dates: First submitted 2024-10-12; First posted 2024-12-05 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Supraventricular Tachycardia (SVtach)
Keywords: Ventricular; Tachycardia
MeSH Terms: conditions — Tachycardia, Supraventricular; Tachycardia | interventions — Adenosine; Verapamil

STUDY DESIGN:
Intervention Model Description: Standard Valsalva maneuver or modified Valsalva maneuver will be attempted on patients according to their allocation of groups. After Three attempts with 5 minutes interval between each attempt if normal sinus rhythm was not achieved. IV pharmacological intervention will made. it includes Injection verapamil 5 mg or adenosine. Each patient will be kept under observation for one hour after normalization of sinus rhythm.
Who Masked: Participant
Masking Description: Modified Valsalva with adenosine will be administered on Monday and Tuesday Conventional Valsalva with adenosine will be administered on Wednesday and Thursday Modified Valsalva with verapamil will be administered on Friday and Saturday
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group A: Conventional Valsalva (Experimental): Performance of forced expiration in the standard manometer tubing to generate a pressure of 40 mmHg for 15 seconds while lying on back or sitting position.
  Interventions: Drug: Adenosine
- Group B: Modified Valsalva Maneuver (Experimental): Patient will be placed in semi-recumbent position and instructed to exhale forcefully in manometer to generate pressure of 40 mmHg for 15 seconds, immediately followed by supine repositioning of the bed, and simultaneous passive leg raising to 45 degree with the help of one assistant standing on the foot side, for 15 seconds.
  Interventions: Drug: Adenosine
- Group C: Modified Valsalva Maneuver (Active Comparator): Patient will be placed in semi-recumbent position and instructed to exhale forcefully in manometer to generate pressure of 40 mmHg for 15 seconds, immediately followed by supine repositioning of the bed, and simultaneous passive leg raising to 45 degree with the help of one assistant standing on the foot side, for 15 seconds.
  Interventions: Drug: Verapamil Injection

INTERVENTIONS:
Drug: Adenosine — Adenosine is a medication belonging to class V antidysrhythmics, used to treat a type of irregular heart rhythm disorder known as paroxysmal supraventricular tachycardia (PSVT)
  Arms: Group A: Conventional Valsalva; Group B: Modified Valsalva Maneuver
Drug: Verapamil Injection — Verapamil is in a class of medications called calcium-channel blockers. It works by relaxing the blood vessels so the heart does not have to pump as hard. It also increases the supply of blood and oxygen to the heart and slows electrical activity in the heart to control the heart rate.
  Other Names: Verapamil
  Arms: Group C: Modified Valsalva Maneuver

SUMMARY:
Supraventricular tachycardia (SVT) is a term widely used to describe tachycardial dysrhythmias, paroxysmal SVT (PSVT) is a narrow term including only AV nodal re-entrant tachycardia (AVNRT) and atrioventricular re-entrant tachycardia (AVRT), both of which can cause discomfort and, in some cases, life-threatening symptoms.

Usually Carotid sinus massage is done to lower the pulse rate and after the standard time specific verapamil dose is administered. In this study after carotid sinus massage Conventional Valsalva or modified Valsalva maneuver will be randomly applied. In case, the normal sinus rhythm (NSR) is not achieved then verapamil of or adenosine dose will be administered to the patients after after taking the consent.

DETAILED DESCRIPTION:
Supraventricular tachycardia (SVT) is a term widely used to describe tachycardial dysrhythmias, paroxysmal SVT (PSVT) is a narrow term including only AV nodal re-entrant tachycardia (AVNRT) and atrioventricular re-entrant tachycardia (AVRT), both of which can cause discomfort and, in some cases, life-threatening symptoms. The incidence of PSVT is approximately 1 in 300 and this prevalence increases with age.

Maneuvers that increase vagus activity have been used to terminate PSVT. Vagal maneuvers reduce the rate of stimulation of the sinus node, slow the rate of delivery to the atrioventricular node, and prolong the refractory period. Vagal-maneuver techniques include carotid sinus massage, the diving reflex, the oculocardiac reflex, and Valsalva maneuvers. Because vagal maneuvers are a non-invasive technique, recent guidelines recommend them as a first-line treatment before medical intervention to terminate PSVT.

Since the 17th century, the Valsalva maneuver (VM) has been used in daily practice and aims to challenge the individual with forced expiration while the glottis is closed, or exhalation to raise the mercury column in tubing of standard manometer to 40 mmHg. In clinical practice, VM has varied success rates (5-20%) in terminating PSVT. It has been found that the patient's posture is an important factor affecting the success of VM. In addition, several studies and case reports have shown that VM with simple, safe modifications (modified VM) is more effective in terminating PSVT. These modifications include pressing the epigastric zone or abdomen for 10 seconds after VM; changing position quickly, such as from being seated to supine; or lifting the feet at a 45-degree angle just after the VM.

Efficacy of SVM in restoring sinus rhythm is less than 25% while of Modified Valsalva maneuver (MVM)) has showed higher efficacy (> 40%).6 However, few studies have evaluated the success rate of modified VM. Therefore, the present randomized controlled study aimed to detect whether modified VM is more effective than standard VM in terminating PSVT.

ELIGIBILITY:
Inclusion Criteria:

* Stable SVT (not requiring cardioversion, fully conscious, maintaining systolic blood pressure of >90mmHg)
* Alert enough and able to give consent
* Able to lie flat and non-painful legs during passive leg raising

Exclusion Criteria:

* Unstable SVT (Semiconscious, drowsy, breathless, systolic BP <90mmHg)
* Not able to give consent
* Orthopnea causing inability to lie flat
* Atrial fibrillation/atrial flutter
* Recent MI (within last 7 days)
* Ongoing ischemia as indicated by chest pain or ST segment depression/elevation in ECG
* Aortic stenosis
* All trimesters of pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-01-27 (Estimated); Study Completion 2025-02-03 (Estimated)

PRIMARY OUTCOMES:
achieve the normal sinus rhythm | 24 to 36 hours
  As the patient came to ER blood pressure and primary information will be collected by the in-charge nurse. then treatment will be provided in following steps First; carotid message will be done. Supraventricular tachycardia (SVT) reverted to normal sinus rhythm (NSR), And if NSR not achieved, Vagal maneuver as mentioned in methodology will be performed, And if NSR not achieved, Randomly, IV verapamil or adenosine will be injected.
  After achieving NSR the patient will be kept under observation for 30 min after that the patient will be asked to visit the Outpatient department (OPD) in the next working day.

SECONDARY OUTCOMES:
Efficacy of standard or modified vagal maneuver | 10 minutes
  Frequency of the patients achieved NSR after standard or modified maneuver will be analyzed for efficacy.
Efficacy of IV verapamil and IV adenosine | 30 to 60 minutes
  carotid message will be done to revert SVT to NSR, Or/And if NSR not achieved Second; Vagal maneuver will be performed, Or/And if NSR not achieved Third, Randomly, IV verapamil or adenosine will be injected in two phases. After achieving NSR the patient will be kept under observation for 30 min.

CONTACTS AND LOCATIONS:
Overall Officials: Hafiz Abdul Manan Shahid, FCPS, Study Director — Punjab Institute of Cardiology
Locations (1):
- Punjab Institute of Cardiology, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
A unique MRN will be assigned to anonymize the patient data. Study director will be the custodian of the data. generalized results will be presented in the conferences and publications

REFERENCES:
- [Background] Corbacioglu SK, Akinci E, Cevik Y, Aytar H, Oncul MV, Akkan S, Uzunosmanoglu H. Comparing the success rates of standard and modified Valsalva maneuvers to terminate PSVT: A randomized controlled trial. Am J Emerg Med. 2017 Nov;35(11):1662-1665. doi: 10.1016/j.ajem.2017.05.034. Epub 2017 May 22. PMID 28552271
- [Background] Rehorn M, Sacks NC, Emden MR, Healey B, Preib MT, Cyr PL, Pokorney SD. Prevalence and incidence of patients with paroxysmal supraventricular tachycardia in the United States. J Cardiovasc Electrophysiol. 2021 Aug;32(8):2199-2206. doi: 10.1111/jce.15109. Epub 2021 Jun 14. PMID 34028109
- [Background] Page RL, Joglar JA, Caldwell MA, Calkins H, Conti JB, Deal BJ, Estes NA III, Field ME, Goldberger ZD, Hammill SC, Indik JH, Lindsay BD, Olshansky B, Russo AM, Shen WK, Tracy CM, Al-Khatib SM. 2015 ACC/AHA/HRS guideline for the management of adult patients with supraventricular tachycardia: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society. Heart Rhythm. 2016 Apr;13(4):e136-221. doi: 10.1016/j.hrthm.2015.09.019. Epub 2015 Sep 25. No abstract available. PMID 26409100
- [Background] Ceylan E, Ozpolat C, Onur O, Akoglu H, Denizbasi A. Initial and Sustained Response Effects of 3 Vagal Maneuvers in Supraventricular Tachycardia: A Randomized, Clinical Trial. J Emerg Med. 2019 Sep;57(3):299-305. doi: 10.1016/j.jemermed.2019.06.008. Epub 2019 Aug 20. PMID 31443919
- [Background] Appelboam A, Reuben A, Mann C, Gagg J, Ewings P, Barton A, Lobban T, Dayer M, Vickery J, Benger J; REVERT trial collaborators. Postural modification to the standard Valsalva manoeuvre for emergency treatment of supraventricular tachycardias (REVERT): a randomised controlled trial. Lancet. 2015 Oct 31;386(10005):1747-53. doi: 10.1016/S0140-6736(15)61485-4. Epub 2015 Aug 24. PMID 26314489